CLINICAL TRIAL: NCT04256109
Title: Women's Access to Mobile Phones and Willingness to Utilize mHealth Interventions for Oral Health Promotion in Egypt: A Cross-Sectional Study
Brief Title: Women's Access to Mobile Phones and Willingness to Utilize mHealth Interventions for Oral Health Promotion in Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ayman Amin Sharaf, Teaching assistant of public health, Ain Shams University
Other Study IDs: 827
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: eHealth; mHealth; Oral Health
Keywords: eHealth; mHealth; Health promotion; Rural area

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2019, it was reported that there were 27.9 million smart phone users and 93.7 million phone subscribers in Egypt. This means that mHealth (which is the use of mobile phones in delivering health-care and public health services) could be a major asset to delivering oral health education to the secluded rural areas or the more under privileged remote areas in the future. However, in order to employ mHealth effectively, it's essential to estimate the percentage of users who, not only have access to mobile technology, but are also willing to utilize mHealth interventions. It is also of great importance to understand the patients' preferences regarding its use. This is in order to tailor an intervention that satisfies their needs for oral health related services. Therefore the aim of this study is to determine the access of Egyptian women to mobile phones, as well as their willingness to utilize mHealth interventions for oral health promotion.

DETAILED DESCRIPTION:
Dental caries and periodontal diseases contribute greatly to the global burden of oral diseases. Unfortunately, this is more observed in the developing countries. This is mainly attributed to the shortage of oral health personnel that Africa suffers from, which results in oral health services being offered mostly to central and urban areas of Africa.

Women, in particular, suffer from health inequalities. Those inequalities are mainly related to socioeconomic status and the geographic region in which they reside.

A study conducted in Egypt in 2014 underlined the oral health inequalities present within the country. This study emphasized the need for oral health promotion plans which are specially directed towards individuals with low-income. That is to provide health equity in terms of access to oral health-care services and quality treatment for all the Egyptian population.

One way to address this problem is the use of Electronic health or "eHealth". mHealth, which is a subset of eHealth, is the use of mobile phones to deliver health-care services through short messaging services (SMS), smart phone applications and voice calls. Several studies highlighted that mHealth can be an effective tool in delivering public health services in a cost effective way and without any geographic barriers.

The multitasking capabilities of mobile phones provide a great chance for chronic disease prevention and improvement as it offers remote health education. Moreover, it provides the patients with increased care and allows for self-management. Mobile phones can also be used as reminders for medications and appointments and allow for immediate contact between the doctor and the patient. This way, mHealth offers uninterrupted care, close monitoring to the patients and rapid response from the doctors' side, this is of course regarded as a more comfortable approach to the patients.

The challenge still lies in the adoption and acceptance of mHealth by the patients, which is controlled by the user's willingness to utilize this new technology. This problem is even more observed in the developing countries. Although mHealth interventions were previously attempted to improve oral health, none were implemented in Egypt. This is the first study to explore the potential use of mHealth for oral health promotion in Egypt.

Study procedure:

* After a comprehensive literature review using electronic databases (PubMed and Web of Science), studies assessing the accessibility to mobile phones, ability to use mobile phones, willingness to utilize mHealth interventions, usage patterns of mobile phones, preferences regarding mHealth, barriers and motivators for participating in mHealth were identified.
* Using nine similar studies, a structured English language interviewer-administered questionnaire was developed after modifying their original questionnaires to serve the aim of our study and ensure culture appropriateness.
* Forward translation of the English questionnaire into Arabic language was done .
* One well-trained investigator will conduct all interviews.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian women.
* Older than 18 years of age.
* Currently residing in Egypt.
* Mentally and medically fit to participate in the study.

Exclusion Criteria:

* Women who do not consent to participate in the study.
* Women seeking emergency dental treatment.
* Women who do not own or share a mobile phone. Their number will be reported by using a flow chart

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Recruited from the outpatient clinics of Faculty of Dentistry, Ain Shams University and five primary healthcare centers located in Cairo and Giza governorates which are affiliated by Egyptian Ministry of Health.
Sampling Method: Non-Probability Sample
Enrollment: 541 (Estimated)
Dates: Start 2020-01-11 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of women in Egypt who have access to mobile phones. | January 2020-June 2020
  Arabic language interviewer-administered questionnaire
Percentage of women in Egypt who are willing to utilize mHealth interventions for oral health promotion. | January 2020-June 2020
  Arabic language interviewer-administered questionnaire

SECONDARY OUTCOMES:
Mobile phones' usage patterns by women in Egypt. | January 2020-July 2020
  Arabic language interviewer-administered questionnaire
Percentage of different methods preferred by women in Egypt for receiving mHealth services | January 2020-July 2020
  Arabic language interviewer-administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Sharaf, Masters, Principal Investigator — Ain Shams University; Amira Badran, Doctorate, Principal Investigator — Ain Shams University; Reham Abou ElFadl, Doctorate, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mangin D, Parascandalo J, Khudoyarova O, Agarwal G, Bismah V, Orr S. Multimorbidity, eHealth and implications for equity: a cross-sectional survey of patient perspectives on eHealth. BMJ Open. 2019 Feb 12;9(2):e023731. doi: 10.1136/bmjopen-2018-023731. PMID 30760515
- [Background] Yamin F, Kaewkungwal J, Singhasivanon P, Lawpoolsri S. Women's Perceptions of Using Mobile Phones for Maternal and Child Health Support in Afghanistan: Cross-Sectional Survey. JMIR Mhealth Uhealth. 2018 Apr 10;6(4):e76. doi: 10.2196/mhealth.9504. PMID 29636317
- [Background] Treskes RW, Koole M, Kauw D, Winter MM, Monteiro M, Dohmen D, Abu-Hanna A, Schijven MP, Mulder BJ, Bouma BJ, Schuuring MJ. Adults with congenital heart disease: ready for mobile health? Neth Heart J. 2019 Mar;27(3):152-160. doi: 10.1007/s12471-019-1237-2. PMID 30758718
- [Background] James DC, Harville C 2nd, Whitehead N, Stellefson M, Dodani S, Sears C. Willingness of African American Women to Participate in e-Health/m-Health Research. Telemed J E Health. 2016 Mar;22(3):191-7. doi: 10.1089/tmj.2015.0071. Epub 2015 Aug 27. PMID 26313323
- [Background] van den Houten MML, Spruijt S, Fokkenrood HJP, Scheltinga MRM, Teijink JAW. User Preferences for Mobile Health Interventions: A Survey among Intermittent Claudication Patients and Their Physical Therapists. Ann Vasc Surg. 2018 Jan;46:249-256. doi: 10.1016/j.avsg.2017.08.020. Epub 2017 Sep 8. PMID 28893710
- [Background] Cormick G, Ciganda A, Cafferata ML, Ripple MJ, Sosa-Estani S, Buekens P, Belizan JM, Althabe F. Text message interventions for follow up of infants born to mothers positive for Chagas disease in Tucuman, Argentina: a feasibility study. BMC Res Notes. 2015 Sep 29;8:508. doi: 10.1186/s13104-015-1498-9. PMID 26419230
- [Background] James DCS, Harville C 2nd. Smartphone Usage, Social Media Engagement, and Willingness to Participate in mHealth Weight Management Research Among African American Women. Health Educ Behav. 2018 Jun;45(3):315-322. doi: 10.1177/1090198117714020. Epub 2017 Jun 13. PMID 28606004
- [Background] Marhefka SL, Turner D, Lockhart E. Understanding Women's Willingness to Use e-Health for HIV-Related Services: A Novel Application of the Technology Readiness and Acceptance Model to a Highly Stigmatized Medical Condition. Telemed J E Health. 2019 Jun;25(6):511-518. doi: 10.1089/tmj.2018.0066. Epub 2019 Jan 18. PMID 30074862